CLINICAL TRIAL: NCT02292459
Title: A Multicenter, Open Label, Non-controlled Phase 3 Clinical Trial of the Efficacy and the Safety for the Relief of Constipation of Polyethylene Glycol 3350
Brief Title: Efficacy and Safety of Polyethylene Glycol 3350 (PEG 3350) for Relief of Constipation (MK-8114-005)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18128; CL2012-15 (Other: Consumer Health Protocol Number); 8114-005 (Other: Merck)
Record Dates: First submitted 2014-11-12; First posted 2014-11-17 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — Solutions; polyethylene glycol 3350; Polyethylene Glycols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEG 3350 (Experimental): Participants will receive a 17 g oral dose of 1 sachet of PEG 3350 mixed in 120 to 240 mL of water, once a day, for 7 days.
  Interventions: Drug: Polyethylene Glycol 3350 Powder for Solution (PEG 3350)
- PEG 4000 (Active Comparator): Participants will receive a 10 to 20 g oral dose of 1 to 2 sachets of PEG 4000 mixed in 120 to 140 mL of water, once a day, for 7 days.
  Interventions: Drug: Polyethylene Glycol 4000 Powder for Solution (PEG 4000)

INTERVENTIONS:
Drug: Polyethylene Glycol 3350 Powder for Solution (PEG 3350)
  Other Names: VivaLAX
  Arms: PEG 3350
Drug: Polyethylene Glycol 4000 Powder for Solution (PEG 4000)
  Other Names: Forlax
  Arms: PEG 4000

SUMMARY:
The purpose of this study is to evaluate the complete resolution of constipation in participants taking PEG 3350 compared to those taking PEG 4000, based on analysis of the number of bowel movements from self-reported bowel movement (BM) data. The complete resolution of constipation is defined as the elimination of straining or of hard/lumpy stools.

ELIGIBILITY:
Inclusion Criteria:

* meets diagnostic criteria for functional constipation. This includes loose stools that are rarely present without the use of laxatives and 2 or more of the following: straining during at least 25% of defecations; lumpy or hard stools in at least 25% of defecations; sensation of incomplete evacuation for at least 25% of defecations; sensation of anorectal obstruction/blockage for at least 25% of defecations; manual maneuvers to facilitate at least 25% of defecations [e.g., digital evacuation, support of the pelvic floor]; and fewer than 3 defecations per week. Criteria for functional constipation must be fulfilled for last 3 months, with symptom onset at least 6 months prior to diagnosis.
* willing to use study drug for up to 7 days as directed, and must agree to record bowel movements (frequency, consistency, etc.) accurately and consistently in a daily diary, and make 3 clinic visits.
* except for constipation, must be otherwise in good health, as determined by physical exam and medical history.
* agrees not to use any other products (drug, herbal, dietary supplements including fiber, etc.) to treat their constipation during the course of the study.
* agrees not to use any medication known to cause constipation during the course of the study.
* agree to maintain a similar diet from the week prior to randomization through the end of the study.
* females must be either surgically sterile, 2 years post-menopausal, or attest that they are using an acceptable method of contraception (including hormonal birth control, intrauterine device [IUD], double barrier methods, or vasectomized partner).
* females of childbearing potential must have urine pregnancy test (human chorionic gonadotropin [HCG]) that is negative at Baseline.
* must be able to read the diaries in Russian.

Exclusion Criteria: - currently under a doctor's care and treatment for constipation.

* have current constipation episode for more than one week prior to randomization.
* history of chronic constipation due to any underlying cause (inflammatory bowel disease, etc.).
* history of more than 3 months of constipation in the past year.
* have severe abdominal pain as the predominant constipation symptom.
* had with bowel movement in 48 hours prior to randomization.
* have celiac disease or known gluten sensitivity.
* history of colorectal cancer, anal abscess, anal fistula, anal fissure, anal stenosis, gastric retention or obstruction, bowel resection, rectocele, or colostomy.
* have known renal or hepatic insufficiency.
* have gastrointestinal bleeding or acute infection.
* history of alcohol or drug abuse.
* history of psychiatric disorders.
* history of significant ongoing medical problems, including kidney disease, or are scheduled for surgical procedures.
* currently taking or have taken within 7 days of randomization a concomitant medication that causes constipation, including opiates, antidepressants, selective serotonin reuptake inhibitors (SSRIs), antimotility agents, and anticholinergics, etc.
* plan to use laxatives during the treatment period other than the study medication.
* have participated in an investigational clinical, surgical, drug or device study within the past 30 days. (Concurrent skin patch testing of cosmetic or suncare products is allowed.)
* pregnant or lactating.
* allergic to polyethylene glycol or maltodextrin.
* employed or have immediate family members employed by a company that manufactures laxative products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Number of bowel movements per week | Up to 7 days after start of treatment

SECONDARY OUTCOMES:
Time to first bowel movement | Up to 7 days after start of treatment
Number of participants who experience changes in straining and hard or lumpy stools | Up to 7 days after start of treatment
Number of participants who experience changes in stool consistency | Up to 7 days after start of treatment
Number of participants who experience changes in the sensation of stool evacuation | Up to 7 days after start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC